CLINICAL TRIAL: NCT06238115
Title: Prophylactic Administration of Tirofiban for Preventing Thromboembolic Events in Stent-assisted Coiling and Flow Diversion Treatments of Unruptured Intracranial Aneurysms
Brief Title: Tirofiban for Reduction of Thromboembolic Events in Endovascular Unruptured Aneurysm Repair
Acronym: TEAR
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSA2022KY009
Record Dates: First submitted 2024-01-17; First posted 2024-02-02 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2024-03

CONDITIONS: Unruptured Intracranial Aneurysm; Flow Diverter; Stent-assisted Coiling; Thromboembolic Events
MeSH Terms: conditions — Thromboembolism | interventions — Tirofiban; Aspirin; Clopidogrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tirofiban group (Experimental): After femoral artery puncture, initial infusion of 0.4μg/kg body weight/minute over 30 minutes, followed by a continuous infusion of 0.1μg/kg body weight/minute for 24 hours.
  Interventions: Drug: Tirofiban; Drug: aspirin, clopidogrel
- Standard medical care (Placebo Comparator): Routine dual antiplatelet therapy (aspirin 100 mg/day, clopidogrel 75 mg/day)
  Interventions: Drug: aspirin, clopidogrel

INTERVENTIONS:
Drug: Tirofiban — Initial infusion of 0.4μg/kg body weight/minute over 30 minutes, followed by a continuous infusion of 0.1μg/kg body weight/minute for 24 hours.
  Arms: Tirofiban group
Drug: aspirin, clopidogrel — aspirin 100 mg/day, clopidogrel 75 mg/day

SUMMARY:
To explore whether administering tirofiban in stent-assisted coiling/flow diverting treatments for participants with unruptured intracranial aneurysms can reduce new ischemic lesions on postoperative DWI sequences compared to conventional dual antiplatelet therapy.

DETAILED DESCRIPTION:
Participants with stent-assisted coiling/flow diverting for unruptured intracranial aneurysms will be enrolled and randomized into two groups: Tirofiban group-after femoral artery puncture, initial infusion of 0.4μg/kg body weight/minute over 30 minutes, followed by a continuous infusion of 0.1μg/kg body weight/minute for 24 hours. Meanwhile, routine dual antiplatelet therapy (aspirin 100 mg/day, clopidogrel 75 mg/day) will be administered. Placebo group-100 mg/day aspirin and 75 mg/day clopidogrel. The primary effectiveness endpoint is the numbers and volumes of ischemic lesions on diffusion weighted imaging (DWI) within 48 hours after procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-80.
2. Participants with unruptured cerebral aneurysms eligible for stent-assisted coiling or flow diversion devices.
3. Completion of preoperative antiplatelet preparation.
4. Signed informed consent.

Exclusion Criteria:

1. Abnormal platelet count (normal reference is 100-300×10^9/L).
2. Allergy to study drugs and anesthetics.
3. Contradictory to MRI examination.
4. Known history of intracranial tumor, arteriovenous malformation, arteriovenous fistula, venous sinus thrombosis, hereditary cerebral small vessel disease, peripheral hemangioma (e.g., aortic aneurysm, limb vascular aneurysm).
5. Known history of cerebral parenchymal hemorrhage, subarachnoid hemorrhage, cerebral infarction, transient ischemic attack, or gastrointestinal bleeding within 6 months.
6. Clear indications for anticoagulation (presumed cardiac source of embolus, e.g., atrial fibrillation, prosthetic cardiac valves known or suspected endocarditis).
7. Antiplatelet drug (exclude aspirin and clopidogrel) being taken within 72 hours; anticoagulant drug (including heparin or oral anticoagulants) being taken within 10 days;
8. Participants with recurrent aneurysms who have received neurointerventional treatment.
9. Inability to follow endovascular procedures due to anatomical difficulties.
10. Severe renal (creatinine exceeding 1.5 times of the upper limit of normal range) or hepatic (ALT or AST > twice the upper limit of normal range) insufficiency.
11. Severe heart failure (NYHA classes III and IV) or severe arrhythmias, including sick sinus syndrome, severe atrioventricular block, and bradycardia-related syncope.
12. Pregnant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2025-11-09 (Actual)

PRIMARY OUTCOMES:
The volumes of ischemic lesions on diffusion weighted imaging within 48 hours after procedure. | within 48 hours after procedure
The numbers of ischemic lesions on diffusion weighted imaging within 48 hours after procedure. | within 48 hours after procedure

SECONDARY OUTCOMES:
Any new stroke events (ischemic stroke or hemorrhagic stroke) within 48-hour and 30-day after procedure. | at postoperative 48-hour and 30-day
Incidence of ischemic stroke within 48-hour and 30-day after procedure. | at postoperative 48-hour and 30-day
Incidence of transient ischemic attack within 48-hour and 30-day after procedure. | at postoperative 48-hour and 30-day
Incidence of ischemic stroke and transient ischemic attack within 48-hour and 30-day after procedure. | at postoperative 48-hour and 30-day
Disabling stroke within 30-day after procedure. | at postoperative 30-day
  Disabling stroke is defined as modified Rankin Scale score >1. The modified Rankin Scale score ranges from 0 to 6, and the higher the score, the greater the degree of disability.

OTHER OUTCOMES:
Moderate and severe bleeding events according to the GUSTO criteria within 48-hour after procedure. | at postoperative 48-hour
Moderate and severe bleeding events according to the GUSTO criteria within 30-day after procedure. | at postoperative 30-day
All bleeding events (severe/moderate bleeding and intracranial hemorrhage) within 48-hour and 30-day after procedure. | at postoperative 48-hour and 30-day
Symptomatic intracranial hemorrhage according to the ECASSIII criteria within 48-hour and 30-day after procedure. | at postoperative 48-hour and 30-day
Total mortality within 48-hour and 30-day after procedure. | at postoperative 48-hour and 30-day
Adverse events/Severe adverse events reported by investigators within 48-hour and 30-day after procedure. | at postoperative 48-hour and 30-day

CONTACTS AND LOCATIONS:
Overall Officials: Jing Jing, Study Chair — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No